CLINICAL TRIAL: NCT07314580
Title: Clinical, Radiographic, Functional and Psychosocial Evaluation of Premolar Autotransplantation to the Anterior Maxillary Region in Young Patients: An Ambispective Observational Study
Brief Title: Clinical and Radiological Evaluation of Dental Autotransplantation in the Anterior Region in Young Patients
Acronym: YATA
Status: Recruiting | Type: Observational
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, MONTSERRAT MERCADE BELLIDO, Principal Investigator, University of Barcelona
Other Study IDs: 63/2025-V3; 63/2025 (Other: CEIm Universitat de Barcelona)
Record Dates: First submitted 2025-12-04; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Tooth Loss; Tooth Injury
Keywords: autotransplantation; tooth autotransplant; premolar donor tooth; anterior maxilla; young patients; root development; CBCT; digital planning; guided surgery; orthodontics; periodontal healing; pulpal healing; traumatic tooth loss; avulsion injuries; trauma-related anterior tooth loss; Dental autotransplantation; Anterior maxillary tooth loss; tooth root development
MeSH Terms: conditions — Tooth Loss; Tooth Injuries; Fractures, Avulsion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autotransplantation Cohort: Young patients (7-15 years) who received or will receive premolar autotransplantation to replace an anterior maxillary tooth, following an identical standardized surgical, orthodontic, radiographic and follow-up protocol. Includes both retrospective and prospective participants.
  Interventions: Procedure: Premolar Autotransplantation

INTERVENTIONS:
Procedure: Premolar Autotransplantation — Premolar autotransplantation performed using a standardized clinical protocol including digital planning (CBCT and STL models), 3D-printed donor tooth replicas, guided or conventional socket preparation, atraumatic donor extraction, extraoral time under 5 minutes and semirigid splinting. Clinical and radiographic follow-up is performed up to 5 years.
  Other Names: Tooth Autotransplantation; Dental Autotransplantation

SUMMARY:
This study aims to evaluate the clinical, radiographic, functional, and patient-reported outcomes of premolar autotransplantation used to replace anterior maxillary teeth in young patients. The study has an ambispective observational design, including a retrospective cohort (patients treated between December 2019 and December 2025) and a prospective cohort (patients enrolled until December 2028).

Participants aged 7 to 15 years who received or will receive premolar autotransplantation to replace an anterior tooth will be followed clinically and radiographically for up to 5 years. Outcomes include tooth survival, periodontal and pulpal healing, root development, complications, orthodontic interactions, restorative needs, and patient satisfaction. The study seeks to identify prognostic factors and long-term success indicators for dental autotransplantation in growing patients.

DETAILED DESCRIPTION:
Premolar autotransplantation is a biologically favorable treatment option for young patients who have lost an anterior maxillary tooth due to trauma, resorption, or restorative failure. This study evaluates outcomes of autotransplantation combining a retrospective cohort (patients treated from 2019 to 2025) and a prospective cohort (patients recruited until 2028). All procedures follow a standardized clinical protocol including digital planning with CBCT and STL models, 3D-printed donor tooth replicas, guided socket preparation when needed, atraumatic donor extraction, extraoral time under 5 minutes, and semirigid splinting.

Clinical and radiographic follow-ups occur at 1 week, 15 days, 1, 2, 3, 6, 9, and 12 months, and annually up to 5 years. Evaluations include mobility, sensitivity, percussion sound, periodontal measurements, gingival recession, root development (Moorrees stages), pulpal healing, and radiographic signs of complications such as resorption or ankylosis. Digital analysis of soft and hard tissues and esthetic outcomes is performed with STL models and CBCT when indicated.

The study also assesses the influence of orthodontic variables (previous treatment, appliance type, timing of movement after transplantation) and restorative parameters (reconstruction chronology). Patient-reported outcomes include satisfaction, esthetics, function, and oral health-related quality of life using validated questionnaires.

Data from both cohorts are anonymized and analyzed descriptively and comparatively, with multivariable modeling to identify prognostic factors.

Although enrollment is defined at the participant level, outcome measures are assessed at the level of the autotransplanted tooth. Participants may contribute more than one autotransplanted tooth to the analysis.

The study will provide long-term evidence regarding success, survival, complications, and perceived outcomes of premolar autotransplantation in growing patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 7 to 15 years.
* ASA I classification.
* Loss or indication for extraction of a maxillary anterior tooth (teeth 12, 11, 21, or 22) due to trauma, resorption, or restorative reasons.
* Availability of a donor first or second premolar with root development between one-half and complete root length.
* Ability to complete at least 2 years of follow-up.
* Parent/guardian consent and minor assent obtained for prospective cases.

Exclusion Criteria:

* Patients older than 15 years.
* Severe systemic disease.
* Inability or unwillingness to attend scheduled follow-up visits.
* Lack of a suitable donor premolar.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Young patients aged 7 to 15 years requiring replacement of a maxillary anterior tooth with a premolar autotransplantation at Dental Esthetic BCN, an accredited CEIm-UB clinical center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Autotransplanted Teeth with Clinical and Radiographic Success | Up to 5 years
  Number of autotransplanted teeth that fulfill all predefined success criteria at each follow-up visit:
  Absence of ankylosis Absence of progressive root resorption Physiological mobility Normal percussion sound Functional stability Absence of clinical signs of infection Each autotransplanted tooth is considered an independent observational unit. In participants with more than one autotransplanted tooth, each tooth is evaluated separately.

SECONDARY OUTCOMES:
Survival Rate of the Autotransplanted Tooth | Up to 5 years
  Number of autotransplanted teeth remaining in situ without extraction during follow-up.
Root Development Stage of the Autotransplanted Tooth | Up to 5 years
  Root development stage of the autotransplanted tooth assessed radiographically using the Moorrees classification.
Pulpal Healing Status of the Autotransplanted Tooth | Up to 5 years
  Number of autotransplanted teeth presenting pulpal healing, defined as pulp canal obliteration or maintained pulp vitality without signs of necrosis, based on clinical testing and radiographic findings.
Periodontal Probing Depth of the Autotransplanted Tooth | Up to 5 years
  Mean periodontal probing depth (in millimeters) measured at six sites around the autotransplanted tooth.
Gingival Recession of the Autotransplanted Tooth | Up to 5 years
  Gingival recession measured in millimeters from the cemento-enamel junction to the gingival margin at the mid-buccal site of the autotransplanted tooth.
Incidence of Root Resorption | Up to 5 years
  Number of autotransplanted teeth presenting inflammatory or replacement root resorption detected radiographically.
Incidence of Ankylosis | Up to 5 years
  Number of autotransplanted teeth presenting clinical and/or radiographic signs of ankylosis.
Orthodontic Treatment After Autotransplantation | Up to 5 years
  Time (in months) from autotransplantation to initiation of orthodontic tooth movement of the autotransplanted tooth.
Number of Restorative Procedures Performed on the Autotransplanted Tooth | Up to 5 years
  Total number of restorative procedures performed on each autotransplanted tooth during follow-up.
Oral Health-Related Quality of Life (OHIP-14 Score) | Up to 5 years
  Mean score of the Oral Health Impact Profile-14 (OHIP-14) questionnaire. Score range: 0-56. Higher scores indicate worse oral health-related quality of life.
Patient Satisfaction with Esthetic Outcome | Up to 5 years
  Patient-reported satisfaction with dental esthetics measured using a Visual Analog Scale (VAS) from 0 to 10, where higher scores indicate greater satisfaction.

OTHER OUTCOMES:
Change in Alveolar Bone Volume at the Autotransplantation Site | Up to 5 years
  Change in alveolar bone volume (in cubic millimeters, mm³) at the autotransplantation site assessed by CBCT superimposition at baseline and follow-up visits, when imaging is clinically indicated.
Change in Gingival Tissue Volume at the Autotransplantation Site | Up to 5 years
  Change in gingival tissue volume (in cubic millimeters, mm³) assessed by STL model superimposition at baseline and follow-up visits, when digital models are available.

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Mercadé, PhD, Principal Investigator — Dental Esthetic BCN / Universitat de Barcelona; Jordi Cadellans, DDS, Principal Investigator — Dental Esthetic BCN / Universitat de Barcelona
Locations (1):
- Dental Esthetic BCN, Barcelona, Barcelons, Spain

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. This decision is based on European GDPR and Spanish data protection laws (LOPDGDD), as the study involves minors and identifiable clinical and radiographic information. Only aggregated, anonymized results will be published in scientific journals. No external researcher will have access to individual-level data.

REFERENCES:
- See also: Dental Esthetic BCN — http://dentalestheticbcn.com